CLINICAL TRIAL: NCT07302386
Title: The Effects of Exercise Management in Parkinson's Disease
Brief Title: Exercise Management in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Gökçe Kartal, MSc, PT, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 949
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease (PD)
MeSH Terms: conditions — Parkinson Disease | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Management Group (Experimental): The self-management group will perform the exercise programme prescribed by the physical therapist and tailored to the patient's needs via a web-based system twice a week for eight weeks, at a time of their choosing.
  Interventions: Other: Telerehabilitation
- Telerehabilitation Group (Active Comparator): Telerehabilitation group will perform the exercise programme prescribed by the physical therapist and tailored to the patient's needs via a web-based system twice a week for eight weeks.
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — The exercises will consist of stretching, strengthening, balance, and neuromotor exercises that the patient can perform independently at home.

SUMMARY:
The aim of this study is to examine the benefits that individuals with Parkinson's disease will gain from the rehabilitation program by enabling them to manage their exercise times independently using telerehabilitation method.

The main research questions examined in this study are as follows:

* Are the improvements in quality of life, walking speed and changes in functionality parameters achieved by individuals with Parkinson's disease through managing their own exercise plans as effective as those achieved through a supervised exercise programme?
* Is it effective for Parkinson's patients to manage their own exercise plans in improving their adherence to exercise?

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a movement disorder characterized by motor and non-motor symptoms, changes in the patient's balance and gait patterns, and a significant impact on daily living activities. Physical therapy and rehabilitation play a crucial role in managing the symptoms resulting from PD. It is known that early participation in a rehabilitation program significantly improves patients' quality of life.

Patients need to incorporate exercise prescriptions designed specifically for them into their lives and participate in a lifelong exercise program. While integrating these exercises into their lives, patients encounter certain barriers and lose their motivation to exercise. These barriers can include transportation, economic problems, time management, and motor and non-motor symptoms.

Home-based exercises and telerehabilitation methods emerge as solutions for dealing with transportation, economic problems, and time management. These methods can be seen as important aids in helping patients develop the habit of exercising.

Patients diagnosed with Idiopathic Parkinson's Disease who meet the inclusion criteria and agree to participate in the study will be included. The demographic information (age, occupation, height, body weight, etc.) and clinical status (duration of diagnosis, medication dosage, etc.) of all participants will be recorded. The Montreal Cognitive Assessment Scale will be used to determine the cognitive level of patients. The motor assessment of patients will be performed using the Cognitive Parkinson's Disease Assessment Scale III. The Montreal Cognitive Assessment Scale will be used to determine the cognitive level of patients. Functional balance and mobility will be assessed using the Timed Up and Go Test and the 10-meter Walk Test. Repetitive movement performance will be assessed using the 5 Repeat Sit-to-Stand Test, and balance level will be assessed using the Activity-Specific Balance Confidence Scale. Quality of life will be assessed using the Parkinson's Disease Quality of Life Questionnaire. Motivation to exercise and self-assessment will be determined using the Behavioral Modifications to Exercise Scale-2. These assessment criteria will be re-evaluated before and after the exercise program. Patients will be given an exercise diary and asked to keep it throughout the program. The System Usability Scale will be used to evaluate the usability of the website developed for this thesis study.

Participants will be randomly assigned to 2 groups. The control group will complete the exercise program assigned to them continuously via the web-based system. The experimental group will complete the exercise program assigned to them at their preferred time within the same day. Exercise programs will be planned for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Idiopathic Parkinson's Disease by a neurologist according to the UK Parkinson's Disease Association Brain Bank clinical diagnostic criteria
* H&Y Stage I-III
* Montreal Cognitive Assessment Scale MoCA≥21
* Having the necessary technological devices to participate in telerehabilitation
* Being able to walk 100 meters
* Having at least a primary school diploma

Exclusion Criteria:

* Presence of a neurological disorder other than Parkinson's disease
* Presence of any cardiopulmonary or musculoskeletal problem that affects gait and balance
* Receiving Deep Brain Stimulation (DBS) treatment or having undergone DBS surgery in the past
* Presence of vision or hearing problems

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-11-07 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Change in motor impairment | Baseline and the end of the 8 weeks exercise program
  The Unified Parkinson's Disease Rating Scale (UPDRS) is used to determine the symptoms and clinical severity of PD. The UPDRS-III subscore will be used to assess changes in motor impairment.
Change in behavioral regulations in exercise | Baseline and the end of the 8 weeks exercise program
  Behavioral Regulations in Exercise Questionnaire-2 consists of 19 items and five subscales. The subscales consist of external regulation, internalized regulation, defined regulation, internal regulation and lack of motivation. It is a 5-point Likert-type scale scored between 0-4.
Change in lower extremity power and endurance | Baseline and the end of the 8 weeks exercise program
  Five Times Sit to Stand Test will be used to measure repetitive movement performance. The patient will be asked to sit down and stand up 5 times as quickly as possible, and this time will be recorded in seconds.
Change in walking speed | Baseline and the end of the 8 weeks exercise program
  10-Meter Walk Test will be applied to assess walking speed. The first 2 meters of the 14-meter distance are allocated for acceleration, the last 2 meters for deceleration, and the time taken to walk the 10-meter distance is recorded. Walking speed is calculated in meters per second.
Change in mobility | Baseline and the end of the 8 weeks exercise program
  Timed Up and Go Test is used to assess mobility, balance, and risk of falling. The patient is asked to stand up from a chair, walk around a cone 3 meters away, and return to sit on the chair. The total time is recorded using a stopwatch.
Change in body position | Baseline and the end of the 8 weeks exercise program
  Activities-Specific Balance Confidence is a measure that assesses a person's level of confidence in their balance both indoors and outdoors. It consists of 16 different activities and is rated on a scale from no confidence (-0) to complete confidence (-100). A higher score indicates a greater level of confidence in balance.
Change in quality of life | Baseline and the end of the 8 weeks exercise program
  The Parkinson's Disease Quality of Life Questionnaire (PDQ-39) will be used to assess quality of life. It consists of 39 items and is composed of 8 sub-parameters: mobility, activities of daily living, stigma, social support, communication, emotional well-being, and physical discomfort. As the score increases, quality of life deteriorates.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Oğuz, PhD, Study Director — Marmara University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franchignoni F, Giordano A, Ronconi G, Rabini A, Ferriero G. Rasch validation of the Activities-specific Balance Confidence Scale and its short versions in patients with Parkinson's disease. J Rehabil Med. 2014 Jun;46(6):532-9. doi: 10.2340/16501977-1808. PMID 24687205
- [Background] Huang SL, Hsieh CL, Wu RM, Tai CH, Lin CH, Lu WS. Minimal detectable change of the timed "up & go" test and the dynamic gait index in people with Parkinson disease. Phys Ther. 2011 Jan;91(1):114-21. doi: 10.2522/ptj.20090126. Epub 2010 Oct 14. PMID 20947672
- [Background] Dean CM, Richards CL, Malouin F. Walking speed over 10 metres overestimates locomotor capacity after stroke. Clin Rehabil. 2001 Aug;15(4):415-21. doi: 10.1191/026921501678310216. PMID 11518442
- [Background] Duncan RP, Leddy AL, Earhart GM. Five times sit-to-stand test performance in Parkinson's disease. Arch Phys Med Rehabil. 2011 Sep;92(9):1431-6. doi: 10.1016/j.apmr.2011.04.008. PMID 21878213
- [Background] Goetz CG, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stebbins GT, Stern MB, Tilley BC, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, Van Hilten JJ, LaPelle N. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Process, format, and clinimetric testing plan. Mov Disord. 2007 Jan;22(1):41-7. doi: 10.1002/mds.21198. PMID 17115387
- [Background] Fahn S. Unified Parkinson's disease rating scale. Recent developments in Parkinson's disease. 1987:153-63.
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468